CLINICAL TRIAL: NCT04310982
Title: The Reliability of a Wearable Inertial System (G-walk) on Gait and Jump Assessment in Healthy Adults.
Brief Title: The Reliability of a Wearable Inertial System in Healthy Adults.
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Gokhan Yazici, Principal Investigator, Gazi University
Other Study IDs: Gazi U
Record Dates: First submitted 2020-03-10; First posted 2020-03-17 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Healthy; Adult
Keywords: Gait; Jump performance; Wearable inertial system; Reliability
MeSH Terms: interventions — Gait Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Health Adults: Forty-nine healthy participants (30 females, 19 males) completed the test-retest protocol with 7 days between tests. Participants were; 23,58±2,65 years of age, 62,9±10,08 kg of weight and 168,76±8,31 cm of height. Participants included in the study did not have any musculoskeletal, neurological or other pathology potentially affecting their gait and jump performance.
  Interventions: Device: The G-Walk sensor system (G-Walk)

INTERVENTIONS:
Device: The G-Walk sensor system (G-Walk) — The G-Walk is a wireless sensor device which is placed on an elastic belt and worn on the waist of the person being evaluated. The device is placed with the center of the device at the fifth lumbar vertebrae and the patient is completely free to walk, run and jump wearing this device. The gait and jump performance of the participants was assessed with the participants wearing this device two times to investigate the test-retest reliability. The second being 7 days after the first.
  Other Names: Gait Analysis

SUMMARY:
Gait analysis is an effective tool used for a variety of purposes, including assessing neurological diseases, risk of falling, orthopedic disability and progress during rehabilitation.The analysis of gait and jump performance must be applicable in a clinical setting. Thus; it needs to be easy to apply in a variety of life situations.The measurements should be reproducible, stable, accurate, capable of distinguishing between normal and abnormal conditions, and cost-effective. Jump measures can predict injury risks, serve as talent identification, and replicate explosive competitive activities of athletes. Furthermore, the performance in vertical jumping can be associated with neuromuscular fatigue.The purpose of this study was to confirm the test-retest reliability of the G-walk wearable sensor system for gait and jump parameters in healthy adults.

DETAILED DESCRIPTION:
The G-Walk determines spatiotemporal parameters as well as pelvic rotations during gait and allows objective and precise analysis of movements with its wearable inertial sensor. It also enables 3D kinematic analysis of the pelvis, providing a functional analysis of disorders in gait caused by neuromuscular diseases The device is placed on an elastic belt and worn on the waist of the person being evaluated, with the center of the device at the fifth lumbar vertebrae. To ensure correct placement of the device, the L4-L5 intervertebral space was palpated via the posterior superior iliac spines.

After the accelerometer was placed, the participants were asked to walk calmly at normal speed, on a 10 m track, and to return to the starting position.

The values and gait characteristics of acceleration in the anteroposterior and mediolateral axes were transferred to the computer software program.

The tilt of the pelvis in the sagittal plane in the flexion-extension direction, the oblique displacement in the coronal plane, the angles of the rotation of movement in the transverse plane and the symmetry values of the right and left sides are obtained. While the symmetry index ranges from 0 to 100, a value closer to 100 indicates that the gait is more symmetrical Following gait assessment, Countermovement jump, static squat jump and Countermovement jump with arms thrust was measured using the device.

ELIGIBILITY:
Inclusion Criteria:

* Accepting to participate in the study,
* Healthy adults,
* Being 18-35 years old,

Exclusion Criteria:

* having any musculoskeletal, neurological or other pathology potentially affecting their gait and jump performance,
* Refusing to participate in the study,
* Having limited cooperation which prevents participation in the study,

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults, 18-35 years old who do not have any concominant diseases.
Sampling Method: Non-Probability Sample
Enrollment: 49 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Gait Analysis | Reliability of the G-Walk in 7 days
  Gait parameters will be assessed via the G-Walk on two separate occasions. The G-Walk is a device that is worn on the waist via an elastic belt. The G-Walk is built with a triaxial accelerometer 16 bit/axes with multiple sensitivity, a triaxial magnetometer 13 bit and a triaxial gyroscope 16 bit/axes with multiple sensitivity. This hardware is capable of acquiring and transmitting data to a computer through a Bluetooth connection and at the end of each analysis an automatic report containing the gait assessment results is ready to be analyzed.
  Gait symmetry values of the right and left sides are obtained within this report. While the symmetry index ranges from 0 to 100, a value closer to 100 indicates that the gait is more symmetrical.
Jump performance | Reliability of the G-Walk in 7 days
  The jump tests protocols included; counter movement jump , squat jump and counter movement jump with arms thrust. At the end of the jump tests, all kinematic parameters concerning the evaluated jump were provided by the software. T Each participant performed a session of three trials for each of the assessed jumps. The jump with the maximum height was accepted for analysis.

SECONDARY OUTCOMES:
Jump height | Reliability of the G-Walk in 7 days
  The jump tests protocols included; counter movement jump , squat jump and counter movement jump with arms thrust. At the end of the jump tests, the height of the jump was given in centimeters by the software.
Peak speed | Reliability of the G-Walk in 7 days
  The jump tests protocols included; counter movement jump , squat jump and counter movement jump with arms thrust. At the end of the jump tests, the peak speed of the jump was given in meters/second by the software.
Maximum concentric power | Reliability of the G-Walk in 7 days
  The jump tests protocols included; counter movement jump , squat jump and counter movement jump with arms thrust. At the end of the jump tests, the maximum concentric power of the jump was given in Newtons by the software.

CONTACTS AND LOCATIONS:
Overall Officials: Gokhan Yazici, Pt. PhD, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No